CLINICAL TRIAL: NCT03357575
Title: The Comparison of Efficacy and Safety of the Mesenchymal Stem Cells From Adipose and Hyaluronic Acid in the Treatment of Adult Knee Osteoarthritis
Brief Title: The Comparison of Efficacy and Safety of the Mesenchymal Stem Cells From Adipose and Hyaluronic Acid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, yangziyi, arthritis clinic and research center, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PUPH20170912
Record Dates: First submitted 2017-11-25; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; adipose; mesenchymal stem cells
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal Stem Cells from adipose (Experimental): Mesenchymal Stem Cells from adipose will be injected.
  Interventions: Biological: Mesenchymal Stem Cells from adipose
- hyaluronic acid (Active Comparator): Hyaluronic acid will be injectied.
  Interventions: Biological: Hyaluronic Acid

INTERVENTIONS:
Biological: Mesenchymal Stem Cells from adipose — inject mesenchymal Stem Cells from adipose
  Arms: Mesenchymal Stem Cells from adipose
Biological: Hyaluronic Acid — inject hyaluronic acid
  Arms: hyaluronic acid

SUMMARY:
The aim of this study was to evaluate the efficacy and safety of Mesenchymal Stem Cells (MSCs) from adipose anticular injection in comparison with hyaluronic acid anticular injection in the treatment of human knee osteoarthritis(OA).

DETAILED DESCRIPTION:
This is a single-centre, quadruple blined, randomized controlled clinical trials with a total of 14 knee osteoarthrits patients as participants, who will be randomly assigned into experiment group or compare group.Participants in experiment group will receive the treatment of MSCs from adipose anticular injection, while participants in compare group will receive hyaluronic acid. Unexplained local and systemic symptoms as well as visual analog scale pain score, WesternOntario McMasterUniversities (WOMAC) Osteoarthritis Index scorewill be assessed at baseline and 2 years after the injection.

ELIGIBILITY:
Inclusion Criteria:

* K / L score of 2-3;
* chronic knee pain;
* no local or systemic infection;
* without obvious contraindication of the joint puncture from hematology and biochemical tests;
* informed consent.

Exclusion Criteria:

* older than 75 years old or less than 18 years old, or without full capacity for civil conduct;
* HIV, hepatitis virus or syphilis virus infection or their serology is positive;
* BMI index is greater than 30;
* congenital or acquired knee deformity;
* pregnant or lactating women;
* tumor patients;
* immunodeficiency patients;
* intra-articular drug injection history within 3 months;
* participating in other clinical trials;
* other patients who researchers believe are not eligible for inclusion such as suffering from other concomitant diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Unexplained local and systemic symptoms or death | 2 years
  The severity of AE must be recorded and graded according to the CTCAE criteria, and its relationship to therapy must be assessed according to the following definition:①not related: there is evidence that the cause of adverse events is not due to intra-articular injection therapy (such as previous conditions, potential diseases, concurrent diseases); ②related: AE and intra-articular injection are time-related and it is known or suspected that intra-articular injection of drugs can cause the AE; ③it can't be assessed.

SECONDARY OUTCOMES:
VAS score | 2 years
  VAS score decrease 3 points or more
WOMAC score | 2 years
  two or more terms of WOMAC score have improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Ziyi Yang, Principal Investigator — arthritis clinic and research center

IPD SHARING:
Plan to Share IPD: No